CLINICAL TRIAL: NCT02721238
Title: Comparison of Colloid (20% Albumin) Versus Crystalloid (Plasmalyte) for Fluid Resuscitation in Cirrhotics With Sepsis Induced Hypotension.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-03
Record Dates: First submitted 2016-03-01; First posted 2016-03-29 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Cirrhosis With Sepsis
MeSH Terms: interventions — Albumins; Plasmalyte A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resuscitation with 30ml/kg plasmalyte (Active Comparator)
  Interventions: Other: Plasmalyte
- Resuscitation with 20% Albumin (Experimental)
  Interventions: Biological: 20% Albumin

INTERVENTIONS:
Biological: 20% Albumin
  Arms: Resuscitation with 20% Albumin
Other: Plasmalyte
  Arms: Resuscitation with 30ml/kg plasmalyte

SUMMARY:
Consecutive cirrhotics who present to emergency department of Institute of Liver & Biliary Sciences with documented or suspected sepsis induced hypotension will be randomized to receive either human albumin infusion over 3 hours or plasmalyte as per requirement. At admission, all patients will undergo physical examination and baseline investigations to identify site of sepsis. The aim of study is to compare the efficacy of using 20% human albumin versus plasmalyte in resuscitation of the patient that is attainment of mean arterial pressure above 65 mm of Hg at three hour after intervention and sustenance of mean arterial pressure above 65 mm of Hg at 6th hour. The randomized patient will be administered 20% albumin (0.5-1.0 gm/kg) for 3 hours, or plasmalyte at the rate of 30ml/kg. After the intervention changes in MAP (Mean Arterial Pressure), lactate level, urine output, incidence of complications, duration of ventilator, ICU (Intensive Care Unit) stay and mortality after one week will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients of cirrhosis with suspected or documented sepsis with MAP < 65 mm Hg

Exclusion Criteria:

* Age <18 years or > 75 yrs
* Already received colloid or 2 litres of fluid within the first 12 hours of presentation
* Already on vasopressors and/or inotropes
* Patients with Spontaneous Bacterial Peritonitis and serum albumin less then 1.5g/dl
* Patient with structural heart disease
* On maintenance hemodialysis
* Other causes of hypotension
* Pregnant or lactating women
* Patients in need for emergent surgical interventions
* Known chronic obstructive lung disease and congestive heart failure
* A previous adverse reaction to human albumin solution

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-11-03 (Actual); Study Completion 2018-11-03 (Actual)

PRIMARY OUTCOMES:
Reversal of hypotension in both groups | 3 hours
  Reversal is defined as Mean Arterial Pressure (MAP) > 65 mmHg after 3 hours of resuscitation

SECONDARY OUTCOMES:
Mortality in both groups | 7 days
Survival time during the first 28 days | 28 days
Proportion of patients with new organ failures. | 28 days
Duration of mechanical ventilation. | 28 days
Requirement of renal-replacement therapy. | 28 days
  Renal-replacement therapy. is defined as patients who required hemodialysis , SLED (Sustained Low efficiency Dialysis) or CRRT (Continous renal replacement therapy).
The duration of the Intensive Care Unit stay. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr Abhinav Verma, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maiwall R, Kumar A, Pasupuleti SSR, Hidam AK, Tevethia H, Kumar G, Sahney A, Mitra LG, Sarin SK. A randomized-controlled trial comparing 20% albumin to plasmalyte in patients with cirrhosis and sepsis-induced hypotension [ALPS trial]. J Hepatol. 2022 Sep;77(3):670-682. doi: 10.1016/j.jhep.2022.03.043. Epub 2022 Apr 20. PMID 35460725